CLINICAL TRIAL: NCT06013371
Title: PDE4 Inhibition in the Treatment of Seborrheic Dermatitis and Papulopustular Rosacea With PF-07038124
Brief Title: PDE4 Inhibition in Seborrheic Dermatitis and Papulopustular Rosacea
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study ended early because interim analysis showed no significant difference between the active and placebo arms.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Benjamin Ungar, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-23-00464
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Seborrheic Dermatitis; Papulopustular Rosacea
MeSH Terms: conditions — Dermatitis, Seborrheic; Rosacea

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 to either drug or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment will be double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF-07038124 (Experimental): PF-07038124 0.02% ointment once daily for 8 weeks
  Interventions: Drug: PF-07038124
- Placebo (Placebo Comparator): Placebo Ointment
  Interventions: Drug: Placebo Ointment

INTERVENTIONS:
Drug: PF-07038124 — topical PDE4 inhibitor
  Arms: PF-07038124
Drug: Placebo Ointment — matching placebo
  Arms: Placebo

SUMMARY:
This study is a double-blind, vehicle-controlled clinical trial. The study will take place at Icahn School of Medicine at Mount Sinai. The study will include 33-39 adult subjects with moderate-to-severe-Seborrheic dermatitis (SD) as well as 33-39 adult subjects with moderate-to-severe papulopustular rosacea (PPR). Subjects will be randomized 2:1 to receive study drug or placebo.

Enrolled subjects will apply topical PF-07038124 0.02% ointment once daily for 8 weeks. They will return for visits at weeks 4, 8, and 12 following study treatment initiation for repeat clinical assessments, medication reviews, tape-strip, blood and urine sample collections, and monitoring for adverse events.

DETAILED DESCRIPTION:
After providing consent, all subjects will be assessed for study eligibility, which includes a review of the subjects past and current medical conditions, familial medical history and detailed review of past and current medications. Subjects will also undergo a review of past topical treatments/therapies for SD or PPR, and clinical assessments (SD: clinical SD score, IGA, Peak Pruritus Numerical Rating Scale [PP-NRS]; PPR: inflammatory lesion count, IGA, PP-NRS).

Subjects who meet inclusion criteria for eligibility may continue with the Baseline Visit (Week 0) or can be scheduled to return for the Baseline Visit within 28 days of the Screening Visit.

At Baseline/Week 0, subjects will undergo clinical assessments (SD: clinical SD Severity Score, IGA, PP-NRS; PPR: inflammatory lesion count, IGA, PP-NRS), review of concomitant medications, standardized clinical photography, and a Dermatology Life Quality index (DLQI) questionnaire. Subsequent clinical assessments including standardized clinical photography, and questionnaire completion will be performed at follow up visits at Week 4, Week 8, and Week 12. Skin tape-strip samples will be collected for mechanistic studies (described below) at baseline (lesional and non-lesional facial skin), Week 4 (lesional facial skin), Week 8 (lesional facial skin), and Week 12 (lesional facial skin). Additional blood samples will be collected and stored at baseline and at Week 8 (or early termination, whichever is first) for potential future mechanistic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age at the time of signing the informed consent document.
* Subject is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures.
* Subject is able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of SD and baseline IGA ≥ 3 with facial involvement
* OR
* Diagnosis of PPR, baseline IGA ≥ 3, and baseline inflammatory lesion count ≥ 12
* Subject agrees to discontinue all treatments for SD and PPR from screening through study completion aside from the study drug
* Subject is judged to be in otherwise good overall health as judged by the investigator, based on medical history, physical examination, and laboratory testing. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on the study drug and for at least 90 days after the last application of the study drug, male and female participants must be willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

  * Option 1: Any one of the following highly effective contraceptive methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy.
  * OR
  * Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

The female subject's chosen form of contraception must be effective by the time the female subject is enrolled into the study.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* Subjects with other skin diseases that would interfere with the study assessment in the opinion of the investigator.
* Active bacterial, fungal, or viral skin infection within 2 weeks from study initiation.
* Subject has clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other major uncontrolled diseases (e.g., malignancy, TB, thromboembolic events) that will affect the health of the subject during the study, or interfere with the interpretation of study results.
* Subject has previously received treatment with oral or topical PDE4 inhibitors.
* Current other topical treatments (e.g., topical corticosteroids, topical calcineurin inhibitors, topical JAK inhibitors, topical metronidazole, topical minocycline, topical ivermectin, topical azelaic acid, topical brimonidine, topical oxymetazalone, topical antihistamines, topical antibacterials) within 2 weeks of baseline.
* Use of systemic non-biologic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus, oral JAK inhibitors within 4 weeks of study initiation.
* Use of systemic biologic immunosuppressive medications, including, but not limited to inhibitors of IL-17, IL-12/23, or IL-23, TNF inhibitors, dupilumab, and abatacept within 12 weeks of baseline.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Current participation in any other study with a biologic investigational medication within 6 months of baseline, or non-biologic investigational medication within 12 weeks of baseline.
* Subject who is pregnant or breast feeding.
* SD or PPR Baseline IGA < 3; PPR inflammatory lesion count <12; SD with no facial involvement.
* Active hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or positive HIV serology at the time of screening for subjects determined by the investigators to be at high-risk for this disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Number of Subjects reaching Investigator's Global Assessment (IGA) success - Seborrheic dermatitis (SD) | Baseline and Week 8
  IGA success defined as: clear (0) or almost clear (1) and a reduction from baseline of ≥2 points score of 0 or 1 at 8 weeks. Full scale is scored from 0-4, higher score indicates more severe symptoms.
  Clear (0) - Complete clear, no signs of SD
  Almost Clear (1) - Only slight pink color or trace amounts of scaling
  Mild (2) - Pink to red color, or slight
  Moderate (3) - Distinct redness or clearly visible scaling
  Severe (4) - Severe score in erythema or scaling
Percent change in lesion count Papulopustular Rosacea (PPR) | Baseline and Week 8
  Percent change from baseline in inflammation (papule/pustule) lesion count at 8 weeks

SECONDARY OUTCOMES:
Change in SD severity score at 8 weeks | Baseline and 8 weeks
  Change from baseline in each component and overall SD score (composed of erythema, scaling, and pruritus components) at 8 weeks. Each component scored 0-4 (0 = absence, 1 = mild, 2 = moderate, 3 = significant, 4 = severe). Total score from 0-12. Higher score indicates more severe symptoms.
Number of patients with treatment success via IGA in PPR | Baseline and 8 weeks
  IGA success is defined as clear (0) or almost clear (1),and a reduction from baseline of ≥2 points score of 0 or 1 at 8 weeks. Full scale is scored from 0-4, higher score indicates more severe symptoms.
  Clear (0) - No inflammatory lesions present, no erythema
  Almost Clear (1) - Very few, small papules/pustules, very mild erythema present
  Mild (2) - Few small or large papules/pustules, moderate erythema
  Moderate (3) - Several small or large papules/pustules, moderate erythema
  Severe (4) - Numerous small and/or large papules/pustules, severe erythema
Change in Clinical Erythema - PPR | Baseline and 8 weeks
  Change from baseline in clinical erythema assessment at 8 weeks. Full scale is scored from 0-4, higher score indicates more severe symptoms.
  Clear (0) -Clear skin with no signs of erythema
  Almost Clear (1) - Almost clear; slight redness
  Mild (2) - Mild erythema; definite redness
  Moderate (3) - Moderate erythema; marked redness
  Severe (4) - Severe erythema; fiery redness
Change in Patient assessment of erythema - PPR | Baseline and 8 weeks
  Change from baseline in patient severity assessment of erythema at 8 weeks. Full scale is scored from 0-4, higher score indicates more severe symptoms.
  Clear (0) - Clear of unwanted redness
  Almost Clear (1) - Nearly clear of unwanted redness
  Mild (2) - Somewhat more redness than I prefer
  Moderate (3) - More redness than I prefer
  Severe (4 - Completely unacceptable redness
Change in Lesion count - PPR | Baseline, 8 weeks, 12 weeks
  Change from baseline and from 8 weeks in inflammatory (papule/pustule) lesion count at 12 weeks
Change in IGA Score - SD and PPR | Baseline, 4 and 8 weeks
  Change from baseline in IGA score at 4 and 8 weeks. Full scale is scored from 0-4, higher score indicates more severe symptoms.
  SD Clear 0 Complete clear, no signs of SD Almost Clear 1 Only slight pink color or trace amounts of scaling Mild 2 Pink to red color, or slight Moderate 3 Distinct redness or clearly visible scaling Severe 4 Severe score in erythema or scaling Clear (0) - Complete clear, no signs of SD
  PPR Clear 0 No inflammatory lesions present, no erythema Almost Clear 1 Very few, small papules/pustules, very mild erythema present Mild 2 Few small or large papules/pustules, moderate erythema Moderate 3 Several small or large papules/pustules, moderate erythema Severe 4 Numerous small and/or large papules/pustules, severe erythema
Percent change in IGA Score - SD and PPR | Baseline, 4 and 8 weeks
  Percent change from baseline in IGA score at 4 and 8 weeks. Full scale is scored from 0-4, higher score indicates more severe symptoms.
  SD Clear 0 Complete clear, no signs of SD Almost Clear 1 Only slight pink color or trace amounts of scaling Mild 2 Pink to red color, or slight Moderate 3 Distinct redness or clearly visible scaling Severe 4 Severe score in erythema or scaling Clear (0) - Complete clear, no signs of SD
  PPR Clear 0 No inflammatory lesions present, no erythema Almost Clear 1 Very few, small papules/pustules, very mild erythema present Mild 2 Few small or large papules/pustules, moderate erythema Moderate 3 Several small or large papules/pustules, moderate erythema Severe 4 Numerous small and/or large papules/pustules, severe erythema
Change in IGA Score - SD and PPR | Baseline and Week 12
  Change from baseline and from 8 weeks in IGA at 12 weeks (i.e., 4 weeks after treatment cessation). Full scale is scored from 0-4, higher score indicates more severe symptoms.
  SD Clear 0 Complete clear, no signs of SD Almost Clear 1 Only slight pink color or trace amounts of scaling Mild 2 Pink to red color, or slight Moderate 3 Distinct redness or clearly visible scaling Severe 4 Severe score in erythema or scaling Clear (0) - Complete clear, no signs of SD
  PPR Clear 0 No inflammatory lesions present, no erythema Almost Clear 1 Very few, small papules/pustules, very mild erythema present Mild 2 Few small or large papules/pustules, moderate erythema Moderate 3 Several small or large papules/pustules, moderate erythema Severe 4 Numerous small and/or large papules/pustules, severe erythema
Change in Peak Pruritus Numerical Rating Scale (PP-NRS) from Baseline at Week 8 | Baseline and Week 8
  Change from baseline in PP-NRS at 8 weeks On a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', patient rates their itch at the worst moment during the previous 24 hours. Higher score indicates more severe symptoms.
Number of related adverse events | 12 weeks
  Number of adverse events reported throughout the study that are deemed related to study drug.
Frequency of adverse events | 12 weeks
  The frequency at which adverse events that are deemed related to study drug are reported throughout the study.
Severity of Adverse Events | 12 weeks
  Severity will be measured as a category (mild, Moderate, severe) according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ungar, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed as aggregated data

DOCUMENTS (1):
  • Informed Consent Form (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT06013371/ICF_001.pdf